CLINICAL TRIAL: NCT02212379
Title: Dual Therapy Combining Raltegravir With Etravirine Maintains a High Level of Viral Suppression Over 96 Weeks in Long-term Experienced HIV-infected Individuals Over 45 Years on a PI-based Regimen: Results From the Phase II ANRS 163 ETRAL Study
Brief Title: Capacity of the Dual Combination Raltegravir/Etravirine to Maintain Virological Success in HIV-1 Infected Patients of at Least 45 Years of Age- ANRS 163 ETRAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-000828-24; ANRS 163 ETRAL (Other: ANRS)
Record Dates: First submitted 2014-07-30; First posted 2014-08-08 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: HIV-1 Infection
Keywords: Raltegravir; Etravirine; aged, 45 and over; Viral load; Efficacy; Safety
MeSH Terms: interventions — Raltegravir Potassium; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- raltegravir and etravirine (Experimental)
  Interventions: Drug: raltegravir and etravirine

INTERVENTIONS:
Drug: raltegravir and etravirine — Raltegravir (RAL, ISENTRESS®) 400 mg tablets will be administered as one 400 mg oral tablet PO twice daily (800 mg per day) after a meal.
  Etravirine (ETR, INTELENCE®) 200 mg tablets will be administered as one 200 mg oral tablet PO twice daily (400 mg per day) after a meal.

SUMMARY:
This multicenter, international, non randomized (single arm), open, phase II trial aims to evaluate the capacity of the dual combination raltegravir/etravirine to maintain virological success in virologically suppressed HIV-1 infected patients, of at least 45 years of age, switching from a boosted PI-containing regimen. Patients will be followed for 96 weeks. The primary endpoint was the proportion of participants with virological success at 48 weeks. Virological success is defined as the absence of 2 consecutive plasma viral load >50 copies/mL within 2 to 4 weeks apart. The study was designed to show an efficacy >90%, assuming a success rate >95%, with a power of 80% and a 5%type-1 error. A total of 160 individuals was required to achieve the objective. The principal secondary endpoint is the proportion of patients in therapeutic success up to week 48 and 96.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Age ≥ 45 years
* Naïve to integrase inhibitor and etravirine
* At least 6 months of stable antiretroviral therapy (ART) including a boosted protease inhibitor, whatever the number of combined drugs
* HIV-RNA plasma VL ≤ 50 copies/mL during the last 24 months prior to screening visit (Week-6/Week-4), documented by at least 4 time-points with no more than one blip in HIV-RNA plasma viral load between 51 and 200 copies/mL
* HIV-RNA plasma VL ≤ 50 copies/mL at screening visit (Week-6/Week-4)
* A genotype is available (on amplified DNA at Week-6/Week-4 Visit and/or on RNA in the medical history of the patient) and shows a virus sensitive to ETR OR no genotype is available (amplification failure on DNA at Week-6/Week-4 Visit and no genotype in the medical history of the patient), there are no virological failure on NNRTI in the medical history
* CD4+ lymphocytes > 200 cells/mm3
* Creatinine < 2.5 x ULN
* CPK (Creatine Phospho Kinase) < 6 ULN (Upper Limit of Normal)
* AST (Aspartate Aminotransferase), ALT (Alanine Aminotransferase) < 5 ULN
* Hemoglobin > 10 g/dL
* Platelets > 100 000/mm3
* Negative urinary pregnancy test and use of efficient contraception for women of childbearing potential
* For French participants only: subject enrolled in or a beneficiary of a Social Security programme (State Medical Aid or AME is not a Social Security programme), article L1121-11 of the Public health code
* Patients with a coverage from a social health
* Signed informed consent

Exclusion Criteria:

* Previous exposure to raltegravir or etravirine
* Presence of any documented integrase inhibitor mutation on DNA genotype at Week-6/Week-4 and/or on RNA in the medical history of the patient
* Positive hepatitis B HBsAg or Positive HBc Ac and negative HBs Ac
* HIV-2 infection
* Active viral hepatitis C requiring a specific treatment during the 24 months of the trial
* Patient with a history of non-compliance or irregular follow-up
* Initiation of a concomitant anti-hypercholesterolemia (e.g. statins) or antidiabetic treatment within the last 3 months prior the screening visit (Week-6 /Week-4)
* Patient using: Clopidogrel (Plavix®), Prasugrel (Effient®), Ticagrelor (Brilinta®), Ticlopidine (Ticlid®), Flurbiprofen (Antadys® - Cebutid®), Rifampin (Rifampicin® - Rifadin® - RofactMC - Rifater®), Rifapentine (Priftin®), St John's wort, Carbamazepine (Tegretol®), Phenobarbital, Phenytoin (Dilantin®),Avanafil (Stendra™), Triazolam (Halcion®)
* Concomitant treatment using interferon, interleukins or any other immunotherapy or chemotherapy
* Concomitant prophylactic or curative treatment for an opportunistic infection
* All conditions (use of alcohol, drugs, etc.) judged by the investigator to possibly interfere with trial protocol compliance, adherence and/or trial treatment tolerance
* Subjects under judicial protection due to temporarily and slightly diminished mental or physical faculties, or under legal guardianship
* Subjects participating in another clinical trial evaluating different therapies and including an exclusion period that is still in force during the screening phase
* Pregnant women or breastfeeding women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales, Groupe Hospitalier Pitié-Salpêtrière, Paris, France; Jacques Reynes, MD, Study Chair — Département des Maladies Infectieuses et Tropicales Hôpital Gui de Chauliac, CHU de Montpellier France; Dominique Costagliola, PhD, Study Director — Inserm UMR S 1136 Université Pierre et Marie Curie Epidémiologie, stratégies thérapeutiques et virologie cliniques dans l'infection à VIH, Paris, France
Locations (19):
- France (16):
  - Hôpital Avicenne, Bobigny
  - Hôpital Jean Verdier, Bondy
  - Hôpital Saint André, Bordeaux
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Croix Rousse, Lyon
  - Hôpital Sainte marguerite, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Hôtel Dieu, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bretonneau, Tours
- Spain (3):
  - Hospital de Bellvitge, Barcelona
  - Hospital de la santa Creu i San Pau, Barcelona
  - Hospital Clinic, Barcelona

REFERENCES:
- See also: Related Info — http://www.anrs.fr/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January and November 2015, 219 patients from 20 sites were screened and 170 patients were enrolled in the study.
Pre-assignment Details: Five patients did not initiate the trial treatment by their own decision, leaving 165 patients for the analysis.
Period: From Baseline to Week 48
Arm/Group | Raltegravir and Etravirine
Started | 165
Completed | 156
Not Completed | 9
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Period: From Week 48 to Week 96
Arm/Group | Raltegravir and Etravirine
Started | 156
Completed | 152
Not Completed | 4
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [48 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 124
  Sub-saharan Africa | 24
  Others | 17
Transmission group [Count of Participants; unit: Participants]
  Men who have Sex with Men | 66
  Heterosexual | 72
  Others/Unknown | 27
Time since HIV diagnosis [Median (Inter-Quartile Range); unit: years] | 19.8 [12.8 to 24.2]
CDC stage C [Count of Participants; unit: Participants] — number of patients with Prior AIDS event
  Participants | 36
CD4 nadir cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 209 [93 to 286]
Hepatitis C co-infection [Count of Participants; unit: Participants] | 16
Antiretroviral treatment (ART) duration [Median (Inter-Quartile Range); unit: years] | 16.9 [11.1 to 19]
Duration of suppressed HIV viremia (<50 copies/ml), [Median (Inter-Quartile Range); unit: years] | 6.9 [3.4 to 9.3]
Duration of last combined antiretroviral therapy (cART) [Median (Inter-Quartile Range); unit: Months] | 58 [32 to 89]
Antiretroviral treatment daily dosing [Count of Participants; unit: Participants]
  once daily | 120
  twice daily | 45
cART at screening [Count of Participants; unit: Participants]
  2NRTIs + PI/r | 107
  NNRTI + PI/r | 11
  PI/r | 35
  Others | 12
Comorbidities [Count of Participants; unit: Participants]
  Cardiovascular | 8
  Dyslipidemia | 53
  High blood pressure | 45
  Diabetes | 10
Active smoking [Count of Participants; unit: Participants] | 60
Former smokers [Count of Participants; unit: Participants] | 31
Alcohol use (>2 glasses/day) [Count of Participants; unit: Participants] | 14
CD4 cell count at screening [Median (Inter-Quartile Range); unit: cells/mm^3] | 700 [525 to 904]
CD8 cell count at screening [Median (Inter-Quartile Range); unit: cells/mm^3] | 678 [525 to 966]
CD4/CD8 ratio at screening [Median (Inter-Quartile Range); unit: ratio] | 0.94 [0.67 to 1.33]
Total cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 5.4 [4.6 to 6.1]
Non-HDL cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 3.9 [3.4 to 4.6]
LDL cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 3.2 [2.7 to 3.8]
HDL cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 1.3 [1.1 to 1.6]
Triglycerides [Median (Inter-Quartile Range); unit: mmol/L] | 1.3 [1.0 to 2.1]
Triglycerides/HDL ratio [Median (Inter-Quartile Range); unit: ratio] | 1.0 [0.6 to 1.8]
Glycaemia [Median (Inter-Quartile Range); unit: mmol/L] | 5.2 [4.7 to 5.7]
Estimated glomerular filtration rate (eGFR, CKD-EPI method) [Median (Inter-Quartile Range); unit: mL/min/1.73 m^2] | 93.9 [79.2 to 103.2]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 24.3 [22.5 to 26.6]
Waist circumference [Median (Inter-Quartile Range); unit: cm] | 92 [84 to 99]
Hip circumference [Median (Inter-Quartile Range); unit: cm] | 95 [90 to 99]
Waist/Hip ratio [Median (Inter-Quartile Range); unit: ratio] | 0.97 [0.9 to 1.03]
Viruses with mutations that could potentially impact etravirine [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Virological Suppression at Weeks 48 and 96
Description: Virological success is defined as the absence of 2 consecutive plasma viral loads (VL) > 50 copies/mL within 2 to 4 weeks of a dual raltegravir/etravirine regimen.
  The proportion of patients who maintained viral suppression under raltegravir plus etravirine was 99.4% (95% confidence interval (95% CI:95.6 -99.9) at week 48 and 98.7% (95% CI: 95.0 -99.7) at week 96
Time Frame: at week48 and at week 96
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of participant
  at week 48 | 99.4 [95.6 to 99.9]
  at week 96 | 98.7 [95.0 to 99.7]

2. Secondary Outcome: Percentage of Patients With Therapeutic Success at Week 48 and Week 96
Description: Therapeutic success was defined as the absence of virological failure (i.e. 2 consecutive plasma viral loads (VL) > 50 copies/mL within 2 to 4 weeks) and the absence of treatment interruption due to adverse event judged by DSMB as related to the study treatment or procedure
Time Frame: weeks 48 and 96
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of participants
  at week 48 | 95.1 [90.5 to 97.5]
  at week 96 | 92.7 [87.5 to 95.8]

3. Secondary Outcome: Percentage of Patients With Trial Treatment Interruption at Week 48 and Week 96
Time Frame: weeks 48 and 96
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of participant
  at week 48 | 4.3 [1.7 to 8.5]
  at week 96 | 6.1 [2.9 to 10.9]

4. Secondary Outcome: Percentage of Patients With With Grade Virological Failure (HIV-RNA Plasma VL Between 51 and 200 Copies/mL)
Time Frame: weeks 48 and 96
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of participants
  at week 48 | 0 [0 to 2.2]
  at week 96 | 0.6 [0.01 to 3.3]

5. Secondary Outcome: Median Time of Virological Failure
Description: Time between the date of the study treatment initiation and the date of virological failure
Time Frame: week 96
Measure: Median (Full Range); unit: weeks
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
weeks | 96 [1 to 96]

6. Secondary Outcome: Percentage of Patients With High Grade of Virological Failure Defined as HIV RNA > 200 Copies/mL
Time Frame: weeks 48 and 96
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of participants
  week 48 | 0.6 [0.01 to 3.3]
  week 96 | 0 [0 to 2.2]

7. Secondary Outcome: Number of Patients With RAL and/or ETR Resistance Mutations Among Those With Virological Failure
Time Frame: week 96
Measure: Number; unit: participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 2
participants | 1

8. Secondary Outcome: Factors Associated With the Occurrence of Plasma HIV-RNA Viral Load > 50 Copies/mL
Time Frame: week 96
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
hazard ratio
  Age >60 years | 3.7 [1.4 to 10.1]
  >=2 glasses/day alcohol consumption | 11.3 [1.5 to 85.1]

9. Secondary Outcome: Evolution of Total Cell-associated HIV-DNA
Time Frame: from day 0 to week 48 and week 96
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 157
percentage of change
  Change from baseline to week 48 | 0 [-29 to 111]
  Change from baseline to week 96 | 0 [-37 to 45]

10. Secondary Outcome: Evolution of CD4+, CD8+ T Cells Counts and CD4/CD8 Ratio
Time Frame: from day 0 to week 48 and week 96
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of change
  CD4: 0-48 week | 1.1 [-10.9 to 16.6]
  CD8: 0-48 week | -1.8 [-18.7 to 16.6]
  CD4/CD8: 0-48 week | 5.7 [-5.7 to 13.8]
  CD4: 0-96 week | 5.0 [-9.4 to 18.9]
  CD8: 0-96 week | -5.2 [-17.1 to 11.2]
  CD4/CD8: 0-96 week | 7.4 [-2.6 to 21.9]

11. Secondary Outcome: Number of Participants Experiencing Adverse Events and Effects
Description: Number of all clinical and biological adverse events effects. Number of grade 3 or 4 clinical and biological adverse events and effects.
Time Frame: From day 0 to week 48 and week 96
Population: After week 48, only 156 participants remained on the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
Participants
  Any AE: 0-48 week | 154
  Grade 3 or 4 AE: 0-48 week | 15
  Any AE : 48-96: number analyzed (Participants) | 156
  Any AE : 48-96 | 108
  Grade 3 or 4 AE: 48-96: number analyzed (Participants) | 156
  Grade 3 or 4 AE: 48-96 | 11

12. Secondary Outcome: Evolution of Metabolic Parameters (Fasting Triglycerides, Total Cholesterol, HDL-cholesterol, LDL-cholesterol and Fasting Glycemia)
Time Frame: from day 0 to week 96
Population: the number analyzed in one or more rows differs from overall number analyzed due to the Non determined data
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
percentage of change
  fasting triglycerides: number analyzed (Participants) | 163
  fasting triglycerides | -18.8 [-40.2 to 10.4]
  total cholesterol: number analyzed (Participants) | 163
  total cholesterol | -0.5 [-16.3 to 7.6]
  HDL-cholesterol: number analyzed (Participants) | 162
  HDL-cholesterol | 5.4 [-7.1 to 21.6]
  LDL-cholesterol: number analyzed (Participants) | 155
  LDL-cholesterol | -4.3 [-19.2 to 10.2]
  fasting glycemia: number analyzed (Participants) | 163
  fasting glycemia | 0 [-7.0 to 10.0]

13. Secondary Outcome: Evolution of the Calibrated 5-year Framingham Risk Score
Description: The Framingham risk score is expressed as a percentage. Higher scores mean a worse outcome and lower scores mean better outcome.
  Median percent change expressed as median (interquartile range (IQR))
Time Frame: from day 0 to week 48 and at week 96
Population: the number of analyzed participants differs from overall participants due to the Non determined data.
Measure: Median (Inter-Quartile Range); unit: Median percent change as median (IQR)
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 128
Median percent change as median (IQR)
  from D0 to week 48 | 1.0 [-22.9 to 37.7]
  from D0 to week 96 | 9.7 [-21.3 to 45.7]

14. Secondary Outcome: Percent Change of Renal Function
Description: Percent change of the estimated Glomerular Filtration Rate (eGFR) calculated using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration Calculator) formula
Time Frame: from day 0 to week 96
Measure: Median (Inter-Quartile Range); unit: Median percent change, as median (IQR)
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
Median percent change, as median (IQR) | -0.6 [-6.6 to 4.2]

15. Secondary Outcome: Evolution of Body Fat Distribution From Day 0 to W96 (DXA Scan Sub-study, 80 Patients)
Description: Evolution of total fat mass, limb fat and trunk fat from day 0 to week 96
Time Frame: from day 0 to week 96
Population: Five participants were not evaluated at week 96
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 75
percentage of change
  Total fat mass, Kg | 12.2 [-1.0 to 24.2]
  Limb fat, Kg | 11.6 [0.7 to 27.8]
  Trunk fat, Kg | 12.2 [-1.9 to 23.3]

16. Secondary Outcome: Sub-study: Bone Mineral Density
Description: • Evolution of bone mineral density (BMD) measured by DXA scans (DXA scan sub-study, 81 patients)
  * Lumbar spine BMD, mg/cm2
  * Total hip BMD, mg/cm2
Time Frame: from day 0, to week 48 and week 96
Population: The number analyzed in one or more rows differs from overall number analyzed due to the missing data
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 81
percentage of change
  Lumbar spine BMD from D0 to week 48 | 0.7 [-1.1 to 2.8]
  Lumbar spine BMD at week 96: number analyzed (Participants) | 80
  Lumbar spine BMD at week 96 | -1.0 [-2.9 to 1.8]
  Total hip BMD from D0 to week 48: number analyzed (Participants) | 79
  Total hip BMD from D0 to week 48 | 0.6 [-0.9 to 1.9]
  Total hip BMD at week 96: number analyzed (Participants) | 79
  Total hip BMD at week 96 | 0 [-0.8 to 1.3]

17. Secondary Outcome: Percentage of Participants With Detectable Seminal HIV-RNA Viral Load at Week 48
Description: • Assessment of HIV-RNA viral load in human male genital compartment (20 patients) at week 48
Time Frame: week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 20
Participants | 1

18. Secondary Outcome: Inflammatory Parameters
Description: • Evolution of the inflammation markers (IL-6hs, sCD14, sCD163, D-Dimers, IP-10, IgG, CRPus and insulin) on frozen plasma aliquots
Time Frame: from day 0 to week 96
Population: The number analyzed in one or more rows differs from overall number analyzed due to the missing data
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 158
percentage of change
  IL-6: number analyzed (Participants) | 144
  IL-6 | 0.8 [-32.4 to 58.8]
  IP-10 | -8.1 [-23.9 to 16.5]
  sCD163 | 0.7 [-21.0 to 20.5]
  sCD14 | -27 [-38 to -8]
  IgG | 0 [-6.8 to 4.8]
  hsCRP: number analyzed (Participants) | 124
  hsCRP | 0 [-34.2 to 55.9]
  D-Dimer: number analyzed (Participants) | 135
  D-Dimer | 16.5 [-2.6 to 40.7]
  Insulin: number analyzed (Participants) | 145
  Insulin | 4.6 [-16.0 to 42.5]

19. Secondary Outcome: Percentage of Participants Reporting a Very Good or an Excellent Quality of Life at Day 0, Weeks 48 and 96
Time Frame: day 0 and weeks 48 and 96
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
Participants
  day 0 | 63
  week 48 | 78
  week 96 | 77

20. Secondary Outcome: Percentage of Participants Compliant With Treatment Program.
Description: The compliance rate was estimated as the number of pills consumed (recorded using the self-reported 90 questionnaire) divided by the number of pills theoretically consumed, classified as low (80%), medium (80%-95%) or high (95%).
Time Frame: at week 0, week 48, and week 96
Population: Among 165 analyzed participated, 155 filled the baseline self-reported adherence questionnaire, 146 at week 48 and 136 at week 96
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 165
Participants
  low (<80) at W0: number analyzed (Participants) | 155
  low (<80) at W0 | 13
  medium (80-95) at W0: number analyzed (Participants) | 155
  medium (80-95) at W0 | 3
  high (>95) at W0: number analyzed (Participants) | 155
  high (>95) at W0 | 139
  low (<80) at W48: number analyzed (Participants) | 146
  low (<80) at W48 | 7
  medium (80-95) at W48: number analyzed (Participants) | 146
  medium (80-95) at W48 | 16
  high (>95) at W48: number analyzed (Participants) | 146
  high (>95) at W48 | 123
  low (<80) at W96: number analyzed (Participants) | 136
  low (<80) at W96 | 12
  medium (80-95) at W96: number analyzed (Participants) | 136
  medium (80-95) at W96 | 9
  high (>95) at W96: number analyzed (Participants) | 136
  high (>95) at W96 | 115

21. Secondary Outcome: Evolution of the Ovarian Reserve From D0 to W48 Measured by AMH on Frozen Aliquots
Description: We measured the Anti-mullerian Hormone (AMH) level to evaluate the ovarian reserve (from D0 to W48)
Time Frame: from day 0, to week 48
Population: We evaluated the AMH level in 40 women with available samples.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 40
ng/mL
  Reproductive activity: D0: number analyzed (Participants) | 12
  Reproductive activity: D0 | 0.172 [0.075 to 0.290]
  Pre-menopausal: D0: number analyzed (Participants) | 6
  Pre-menopausal: D0 | 0.009 [0.008 to 0.012]
  Post-menopausal: D0: number analyzed (Participants) | 22
  Post-menopausal: D0 | 0.009 [0.008 to 0.0095]
  Reproductive activity: W48: number analyzed (Participants) | 12
  Reproductive activity: W48 | 0.152 [0.034 to 0.400]
  Pre-menopausal: W48: number analyzed (Participants) | 6
  Pre-menopausal: W48 | 0.008 [0.006 to 0.010]
  Post-menopausal: W48: number analyzed (Participants) | 22
  Post-menopausal: W48 | 0.005 [0.004 to 0.007]

22. Secondary Outcome: Evolution of the Level of MCP1 From D0 to W48 on Frozen Samples
Time Frame: from day 0, to week 48
Population: We evaluated the MCP1 level in 40 women with available samples.
Measure: Median (Inter-Quartile Range); unit: Percentage change
Arm/Group | Raltegravir and Etravirine
Number analyzed (Participants) | 40
Percentage change
  Premenopausal with mesurable AMH: number analyzed (Participants) | 12
  Premenopausal with mesurable AMH | 3.1 [-18.9 to 15.3]
  Premenopausal with reduced ovarian reserve: number analyzed (Participants) | 6
  Premenopausal with reduced ovarian reserve | 3.5 [-2.1 to 10.9]
  Post-menopausal: number analyzed (Participants) | 22
  Post-menopausal | -2.4 [-13.7 to 14.2]

23. Secondary Outcome: Sub-study in Women : Comparison of the Metabolic/Inflammatory Profile in Women According to Their Ovarian Reserve and Menopausal Status at D0 and Its Evolution up to Week 96
Description: Metabolic markers measures are total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides.
  Inflammatory and innate immune activation markers measures are: IL-6hs, sCD14, sCD163, D-Dimers, IP-10, IgG, hsCRP and Insulin.
  Ovarian reserve measure is AMH
Time Frame: from day 0, to week 96
Population: We evaluated the AMH level in 40 women with available samples
Measure: Median (Inter-Quartile Range); unit: Percentage of change
Groups:
- Premenopausal With Mesurable AMH: AMH was detectable (level >0.06 ng/ml) indicating that they had an ovarian reserve and a status of reproductive activity
- Premenopausal With Reduced Ovarian Reserve: AMH<0.02 ng/ml at inclusion in non-menopausal women who were classified as pre-menopausal
- Postmenopausal: The menopausal status was recorded by the questionnaire at inclusion
Arm/Group | Premenopausal With Mesurable AMH | Premenopausal With Reduced Ovarian Reserve | Postmenopausal
Number analyzed (Participants) | 12 | 6 | 22
Percentage of change
  Total cholesterol | 6.62 [-7.99 to 15.88] | 6.91 [2.38 to 17.77] | -11.35 [-15.81 to 2.38]
  LDL-cholesterol | 5.52 [-20.13 to 27.13] | 5.62 [-13.10 to 22.08] | -6.58 [-19.77 to -0.07]
  HDL-cholesterol | 18.47 [3.90 to 27.79] | 27.74 [16.77 to 42.86] | -4.84 [-11.35 to 9.92]
  Triglycerides | 5.59 [-28.10 to 27.57] | -38.37 [-45.18 to -13.70] | -0.99 [-33.12 to 16.67]
  sCD14 | -31.6 [-39.2 to -5.4] | -32.8 [-43.2 to -23.4] | -18.8 [-36.5 to -3.6]
  sCD163 | 10.8 [-9.7 to 32.3] | 15.9 [-9.2 to 34.2] | 4.8 [-21.0 to 49.0]
  hsCRP | 5.7 [-36.0 to 31.5] | 31.8 [-63.3 to 122.6] | -31.4 [-44.7 to 19.0]
  D-dimers: number analyzed (Participants) | 10 | 5 | 19
  D-dimers | 6.8 [-18.3 to 27.2] | 34.8 [14.6 to 90.2] | 23.1 [-7.9 to 46.9]
  IgG | 0.7 [-5.3 to 3.7] | 1.8 [-9.9 to 4.2] | -1.2 [-7.8 to 3.4]
  IL-6hs: number analyzed (Participants) | 12 | 5 | 20
  IL-6hs | 5.9 [-21.6 to 62.7] | -49.9 [-50.5 to -20.8] | -0.9 [-40.7 to 38.9]
  IP-10 | -18.3 [-37.3 to -2.9] | 8.2 [-8.2 to 33.1] | -5.4 [-34.9 to 31.1]
  Insulin: number analyzed (Participants) | 12 | 6 | 21
  Insulin | -29.2 [-48.6 to -0.4] | 30.3 [-7.9 to 50.0] | 11.4 [-14.0 to 32.8]

24. Secondary Outcome: Sub-study in Women : Comparison of the Evolution Fat Distribution Measured by DXA Scan and Body Weight According to AMH Status
Description: BMI, Hip circumference, Waist circumference, waist/hip ratio, Limb fat, Trunk fat, Total fat, Limb lean, Trunk lean, and Total lean
Time Frame: from day 0, to week 96
Population: AMH level were evaluated in 40 women with available samples
Measure: Median (Inter-Quartile Range); unit: Percentage of change
Arm/Group | Premenopausal With Mesurable AMH | Premenopausal With Reduced Ovarian Reserve | Postmenopausal
Number analyzed (Participants) | 12 | 6 | 22
Percentage of change
  Body mass index (BMI) | -0.96 [-5.49 to 2.59] | 5.69 [0.00 to 12.20] | 2.07 [-1.10 to 5.17]
  Hip circumference: number analyzed (Participants) | 7 | 6 | 17
  Hip circumference | 7.06 [-3.64 to 11.71] | 2.80 [-1.16 to 8.85] | 3.09 [-0.94 to 6.19]
  Waist circumference: number analyzed (Participants) | 7 | 6 | 17
  Waist circumference | 2.74 [-4.76 to 6.54] | 4.20 [2.80 to 15.85] | 6.52 [1.11 to 8.20]
  Waist/hip ratio: number analyzed (Participants) | 7 | 6 | 17
  Waist/hip ratio | -3.43 [-4.63 to -1.17] | 0.02 [-1.42 to 10.54] | 1.85 [-1.17 to 5.29]
  Limb fat: number analyzed (Participants) | 5 | 3 | 9
  Limb fat | -2.94 [-5.84 to 1.94] | 6.74 [-1.62 to 16.91] | 10.89 [-0.03 to 28.22]
  Trunk fat: number analyzed (Participants) | 5 | 3 | 9
  Trunk fat | -6.90 [-12.91 to -2.27] | 18.80 [10.32 to 25.31] | 21.27 [5.96 to 39.40]
  Total fat: number analyzed (Participants) | 5 | 3 | 9
  Total fat | -2.59 [-8.93 to -2.13] | 16.77 [7.35 to 17.91] | 24.39 [0.61 to 31.63]
  Limb lean: number analyzed (Participants) | 5 | 3 | 9
  Limb lean | -0.70 [-1.89 to 0.96] | 2.13 [-2.73 to 6.21] | -1.44 [-2.91 to 1.93]
  Trunk lean: number analyzed (Participants) | 5 | 3 | 9
  Trunk lean | -0.79 [-4.60 to 2.54] | 5.53 [1.93 to 20.75] | -3.24 [-6.20 to -0.34]
  Total lean: number analyzed (Participants) | 5 | 3 | 9
  Total lean | -1.35 [-1.93 to 1.14] | 5.83 [2.02 to 8.12] | -3.01 [-4.14 to 2.94]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from baseline to week 48 and 96
Arm/Group | Raltegravir and Etravirine
All-Cause Mortality (participants affected / at risk) | 0/165
Serious Adverse Events (participants affected / at risk) | 26/165
Other Adverse Events (participants affected / at risk) | 23/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir and Etravirine (N=165)
Prostatitis (Reproductive system and breast disorders) | 3 (3)
Stroke (Nervous system disorders) | 2 (2)
Hospitalization further diagnosis (Investigations) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Delirious (Nervous system disorders) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Loss of teeth (General disorders) | 1 (1)
Open wound of back (General disorders) | 1 (1)
Osteoarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Parotidectomy (Surgical and medical procedures) | 1 (1)
Post herpetic neuralgia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Anal abcess (Infections and infestations) | 1 (1)
AST increased (Hepatobiliary disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbago (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pulmonary carcinomia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir and Etravirine (N=165)
Headache (Nervous system disorders) | 6 (7)
Asthenia (Nervous system disorders) | 4 (4)
Insomnia (Nervous system disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Drowsiness (Nervous system disorders) | 2 (2)
dysgeusia (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The absence of a comparator arm, which in terms of impact on fat, bone density and inflammation/activation markers may limit the interpretation of the observed changes over time. One limitation is the small number of women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study protocol, Statistical Analysis (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02212379/Prot_SAP_ICF_000.pdf
  • Informed Consent Form: Informed Consent Form (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT02212379/ICF_001.pdf